CLINICAL TRIAL: NCT02524509
Title: An Inverstigational Clinical Trial for the Safety and Efficacy Evaluation of Chondron(Autologous Cultured Chondrocyte)Compared With Mircrofracture Surgery in Subjects With Cartilage Defects of the Knee Joint
Brief Title: the Safety and Efficacy Evaluation of Chondron Compared With Mircrofracture of Knee
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07CON
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Defect of Articular Cartilage; Articular Cartilage Disorder of Knee; Degeneration; Articular Cartilage, Knee
Keywords: Chonodron; Microfracture; autologous cultured chondrocyte; cartilage defect of knee
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CHONDRON: Patients who already received autologous chondrocyte implantation using CHONDRON (Autologous Cultured Chondrocyte) for knee cartilage defects
- Microfracture: patients already underwent microfracture

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of Chondron(autologous cultured Chondrocyte) by comparing between Chondron implantation and Microfracture.

DETAILED DESCRIPTION:
It is an open clinical trial. Among the patients who received autologous cartilage cell graft using CHONDRON (autologous cartilage cells) in the past (investigational group) or microfracture (control group), the subjects who agreed to participate in the trial voluntarily will undergo the screening process that assesses the suitability of the subjects to the clinical trial and participate in the clinical trial. During the clinical trial period, the subjects should follow the instruction of clinician in charge. Hospital visit is total 2 times* regularly. At the visit, to evaluate the efficacy according to the protocol, the subject will be examined by clinicians, MRI test, and X-ray. If the selection time and the visit time are same, hospital visit will be one time*.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients who underwent autologous chondrocyte implantation using CHONDRON (autologous cultured chondrocyte) or patients underwent microfracture more than 2 years ago.

2. Patients who meet the above criteria 1, the patient or a guardian agreed to participate in the clinical trial, and signed a written agreement form

Exclusion Criteria:

- 1. Patients with psychological disease or other patients who are determined to be unsuitable to this clinical trial by the investigators conducting the clinical trial.

2. Patients who underwent autologous chondrocyte implantation applying CHONDRON (autologous cultured chondrocyte) or microfracture, and the lesion was treated with other procedures subsequently.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Total 50 patients. Patients who received autologous chondrocyte implantation using CHONDRON (autologous cultured chondrocyte) for knee osteoarthritis or patients underwent microfracture. There are total 28 patients who get CHONDRON grafting until now. Considering dropout rate, the selected number of investigational group is total 25, and 25 of equivalent control group is planned.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Score change of KOOS(Knee Injury and Osteoarthritis Outcome) | Screening, post op 2years
  comparison of the difference between a group with Chondron Implantation and a group with Microfracture.

SECONDARY OUTCOMES:
Score change of 100 Vas(visual Analog System) | Screening, post op 2years
  Comparison the difference between a group with Chondron Implantation and a group with Microfracture
Score change of IKDC (International Knee Documentation Committee) | screening, post op 2 years
  comparison the difference between a group with Chondron Implantation and a group with Microfracture
Score change of KSS(Knee Society Score) | Screening, Post op 2 years
  Comparision the difference between a group with Chondron Implantation and a group with Microfracture.
Comparing MRI results | Screening, Post op 2years
  Comparison the difference of morphological improvement from MRI image between a group with Chondron Implantation and a group with Microfracture

CONTACTS AND LOCATIONS:
Overall Officials: Myung Goo Kim, MD, Principal Investigator — Inha University Medical School Hospital
Locations (1):
- Inha University Medical School Hospital, Incheon, Inchoen, South Korea